CLINICAL TRIAL: NCT03712410
Title: A Problem Solving Intervention for Hospice Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Demiris, PhD (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor-Investigator, George Demiris, PhD, PIK Professor, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 828990; R01NR012213 (NIH)
Record Dates: First submitted 2018-10-15; First posted 2018-10-19 (Actual); Results first posted 2023-01-25 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-01

CONDITIONS: Anxiety Generalized; Quality of Life; Depression
MeSH Terms: conditions — Generalized Anxiety Disorder; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (PISCES face to face) (Active Comparator): Family caregivers will receive three sessions of the PISCES intervention in person. The agenda for the first face to face visit for caregivers (suggested timeline 5-7 days after hospice admission) includes an explanation of the purpose of the visit/call. During the first session, the interventionist works on steps one and two of the ADAPT model, namely "Attitude" and "Defining the Problem and Setting Realistic Goals." During the second visit (suggested timeline 11-13 days after hospice admission) the interventionist covers steps three and four of the ADAPT model. Step three encourages caregivers in being creative and generating alternative solutions. Step four focuses on predicting the consequences and developing a solution plan. The third visit (suggested timeline 16-18 days after hospice admission) focuses on step five, namely trying out the solution plan and determining if it works.
  Interventions: Behavioral: PISCES
- Group 2 (PISCES delivered in a hybrid format) (Experimental): In this group, participants will receive the PISCES intervention in three sessions; however, the first session will be delivered face to face and the other two via video. The three intervention sessions will be scheduled with a suggested timeline between days 5 and 18 of the hospice admission. The first session will take place in person (suggested timeline 5-7 days after hospice admission). After the first session where the in-person encounter will allow for the establishment of rapport between the interventionist and the caregiver, the second session (suggested timeline 11-13 days after hospice admission) and the third session (suggested timeline 16-18 days after hospice admissions) will be conducted via live videoconferencing. If the caregiver already has access to a computer and Internet, they will utilize the videoconferencing solution. If videoconferencing is not feasible, the sessions will be delivered over the regular phone.
  Interventions: Behavioral: PISCES
- Group 3 (PISCESplus) (Experimental): PISCESplus is meant to be an enhanced version of the PISCES intervention including the original problem solving therapy modules with the addition of positive reappraisal elements. The suggested timeline for the first session which will be in person is 5-7 days after hospice admission. At the end of the first session, the interventionist will ask the caregiver to take the time to think about and identify some positive aspects of caregiving.
  At the end of the second session (which is scheduled to take place via video approx. 11-13 days after admission) the interventionist will ask the caregiver to go over the benefits or positive aspects of caregiving that they had identified and ask them to comment as to why they perceive these as positive or beneficial.
  The third session will also take place via video.
  Interventions: Behavioral: PISCES
- Group 4 (PISCESplus online) (Experimental): Participants in this group receive the PISCES plus intervention (the PISCES intervention with the enhancement of the positive reappraisal elements) delivered fully online. All assessments and sessions take place online.
  Interventions: Behavioral: PISCES

INTERVENTIONS:
Behavioral: PISCES — The intervention is based on Problem Solving Therapy and is a coping skills intervention designed for family caregivers of hospice patients.

SUMMARY:
Hospice care is conceptualized as quality compassionate care for people facing a life-limiting illness, with services that cover clinical care, pain management, and emotional and spiritual support tailored to patients' and families' needs and preferences. Family members, spouses, friends or others who assume the unpaid or informal caregiving role are essential to the delivery of hospice services; however, stress and caregiver burden can negatively affect caregivers' morbidity and mortality. The emotional needs of individuals caring for dying persons at home are not well attended, and interventions aiming to provide support to hospice caregivers are notably lacking. The investigator team recently completed a study with 514 hospice caregivers to test a problem-solving therapy (PST) intervention tailored specifically for the hospice setting, entitled PISCES (Problem-solving Intervention to Support Caregivers in End of Life care Settings). The findings demonstrate that the PISCES intervention when delivered face to face was effective leading to statistically significant decrease in anxiety and increase in quality of life when compared to the other groups (video group and attention control). An additional lesson learned from that RCT study was that caregivers wanted to focus not only on specific problems or challenges, but also on recognizing the positive aspects of caregiving. This approach of positive reappraisal has been found to enhance problem solving interventions in other settings. The specific aims of this new study are: 1) to compare the effectiveness of the PISCES intervention when delivered face to face and when delivered in a hybrid platform (with the first session in person and remaining sessions via video) to hospice caregivers; 2) to compare the effectiveness of the PISCES intervention to the refined PISCES intervention (PISCESplus) that integrates positive reappraisal elements; 3) to assess caregivers' perceptions of and satisfaction with the PISCESplus intervention; and 4) to conduct a cost analysis of the three intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* enrolled as a family/informal caregiver of a hospice patient
* 18 years or older
* with access to a standard phone line or Internet and computer access at home
* without functional hearing loss or with a hearing aid that allows the participant to conduct telephone conversations as assessed by the research staff (by questioning and observing the caregiver)
* speak and read English, with at least a 6th-grade education

Exclusion Criteria:

* hearing or visual impairment that prohibits from conducting phone conversations or video conference sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The investigator's inclusion criteria cover all genders (and gender is based on self-representation of gender identity).
Enrollment: 523 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Demiris, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 (PISCES-f2f): Family caregivers will receive three sessions of the PISCES intervention in person. The agenda for the first face to face visit for caregivers (suggested timeline 5-7 days after hospice admission) includes an explanation of the purpose of the visit/call. During the first session, the interventionist works on steps one and two of the ADAPT model, namely "Attitude" and "Defining the Problem and Setting Realistic Goals." During the second visit (suggested timeline 11-13 days after hospice admission) the interventionist covers steps three and four of the ADAPT model. Step three encourages caregivers in being creative and generating alternative solutions. Step four focuses on predicting the consequences and developing a solution plan. The third visit (suggested timeline 16-18 days after hospice admission) focuses on step five, namely trying out the solution plan and determining if it works.
  PISCES: The intervention is based on Problem Solving Therapy and is a coping skills intervention designed for family caregivers of hospice patients.
- Group 2 (PISCES Video): In this group, participants will receive the PISCES intervention in three sessions; however, the first session will be delivered face to face and the other two via video or phone. The three intervention sessions will be scheduled with a suggested timeline between days 5 and 18 of the hospice admission. The first session will take place in person (suggested timeline 5-7 days after hospice admission). After the first session where the in-person encounter will allow for the establishment of rapport between the interventionist and the caregiver, the second session (suggested timeline 11-13 days after hospice admission) and the third session (suggested timeline 16-18 days after hospice admissions) will be conducted via live videoconferencing. If the caregiver already has access to a computer and Internet, they will utilize the videoconferencing solution. If videoconferencing is not feasible, the sessions will be delivered over the regular phone.
  PISCES: The intervention is based on Problem Solving Therapy and is a coping skills intervention designed for family caregivers of hospice patients.
- Group 3 (PISCESplus): PISCESplus is meant to be an enhanced version of the PISCES intervention including the original problem solving therapy modules with the addition of positive reappraisal elements. The suggested timeline for the first session which will be in person is 5-7 days after hospice admission. At the end of the first session, the interventionist will ask the caregiver to take the time to think about and identify some positive aspects of caregiving.
  At the end of the second session (which is scheduled to take place via video approx. 11-13 days after admission) the interventionist will ask the caregiver to go over the benefits or positive aspects of caregiving that they had identified and ask them to comment as to why they perceive these as positive or beneficial.
  The third session will also take place via video.
  PISCES: The intervention is based on Problem Solving Therapy and is a coping skills intervention designed for family caregivers of hospice patients.
- Group 4 PISCESplus Online: In this group, participants receive the entire intervention (PISCES plus-so the PISCES intervention with the positive reappraisal enhancements) online and complete all surveys electronically. All pre-and post assessments are conducted online and the PISCES sessions are carried out online as well.
Period: Overall Study
Arm/Group | Group 1 (PISCES-f2f) | Group 2 (PISCES Video) | Group 3 (PISCESplus) | Group 4 PISCESplus Online
Started | 154 | 152 | 154 | 63
Completed | 115 | 106 | 101 | 46
Not Completed | 39 | 46 | 53 | 17

BASELINE CHARACTERISTICS:
Population: Participants were randomly assigned to each of these groups. They reported baseline demographics upon consenting to participate in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (PISCES-f2f) | Group 2 (PISCES Video) | Group 3 (PISCESplus) | Group 4 PISCESplus Online | Total
Number analyzed (Participants) | 154 | 152 | 154 | 63 | 523
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (12.7) | 58.8 (12.8) | 57.4 (12.2) | 56.1 (17.2) | 57.4 (13.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 23 | 34 | 20 | 12 | 89
  Female | 129 | 113 | 130 | 51 | 423
  Unknown or Decline to Answer | 2 | 5 | 4 | 0 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 11 | 9 | 35
  Not Hispanic or Latino | 138 | 136 | 134 | 51 | 459
  Unknown or Not Reported | 9 | 8 | 9 | 3 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 2
  Asian | 3 | 1 | 3 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 64 | 56 | 53 | 23 | 196
  White | 72 | 82 | 79 | 28 | 261
  More than one race | 12 | 8 | 14 | 8 | 42
  Unknown or Not Reported | 3 | 5 | 4 | 1 | 13
Caregiver Generalized Anxiety Disorder (GAD-7) Score [Mean (Standard Deviation); unit: units on a scale] | 6.69 (5.4) | 5.74 (4.9) | 6.32 (4.9) | 5.85 (5.2) | 6.2 (5.1)
Caregiver PHQ-9 Score [Mean (Standard Deviation); unit: units on a scale] | 7.54 (5.7) | 6.6 (5.4) | 6.99 (5.3) | 6.78 (5.36) | 7.0 (5.5)
Caregiver Quality of Life Index (CQLI-R) [Mean (Standard Deviation); unit: units on a scale] | 27.7 (8.0) | 28.5 (8.4) | 29.32 (7.2) | 28.31 (7.7) | 28.5 (7.9)
Caregiver Status [Count of Participants; unit: Participants]
  Bereaved | 43 | 47 | 46 | 4 | 140
  Active | 107 | 102 | 103 | 59 | 371
  Unknown or Not Reported | 4 | 3 | 5 | 0 | 12
Caregiver Diagnosis [Count of Participants; unit: Participants]
  Cancer | 11 | 6 | 10 | 5 | 32
  Dementia | 2 | 3 | 2 | 13 | 20
  Other | 38 | 35 | 33 | 5 | 111
  Unknown or Not Reported | 103 | 108 | 109 | 40 | 360
Caregiver Dementia [Count of Participants; unit: Participants]
  No | 14 | 8 | 9 | 1 | 32
  Yes | 6 | 4 | 5 | 21 | 36
  Don't Know | 35 | 35 | 35 | 5 | 110
  Unknown or Not Reported | 99 | 105 | 105 | 36 | 345
Caregiver Marital Status [Count of Participants; unit: Participants]
  Single/Never Married/Partnered | 37 | 38 | 25 | 20 | 120
  Married/Partnered | 67 | 69 | 76 | 33 | 245
  Widowed | 23 | 16 | 20 | 2 | 61
  Separated/Divorced | 18 | 18 | 14 | 7 | 57
  Decline to Answer | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 9 | 10 | 19 | 1 | 39
Caregiver Education [Count of Participants; unit: Participants]
  Less than High School | 2 | 1 | 2 | 0 | 5
  High School/GED | 24 | 27 | 25 | 6 | 82
  Some College/Associate Degree | 38 | 42 | 43 | 17 | 140
  Bachelor's Degree | 40 | 27 | 37 | 17 | 121
  Graduate/Professional Degree | 41 | 45 | 28 | 22 | 136
  Unknown or Not Reported | 9 | 10 | 19 | 1 | 39
Caregiver Relation [Count of Participants; unit: Participants]
  Spouse/Partner | 41 | 42 | 41 | 15 | 139
  Adult Child | 70 | 69 | 74 | 38 | 251
  Parent | 7 | 7 | 5 | 1 | 20
  Sibling | 6 | 4 | 3 | 1 | 14
  Other | 20 | 20 | 12 | 7 | 59
  Decline to Answer | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 9 | 10 | 19 | 1 | 39
Care Receiver Gender [Count of Participants; unit: Participants]
  Male | 69 | 59 | 69 | 15 | 212
  Female | 75 | 83 | 64 | 47 | 269
  Unknown or Not Reported | 10 | 10 | 21 | 1 | 42
Care Receiver Ethnicity [Count of Participants; unit: Participants]
  Hispanic | 6 | 8 | 11 | 5 | 30
  Non-Hispanic | 136 | 133 | 120 | 55 | 444
  Decline to Answer | 2 | 1 | 2 | 2 | 7
  Unknown or Not Reported | 10 | 10 | 21 | 1 | 42
Care Receiver Race [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 5 | 2 | 3 | 3 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 63 | 55 | 50 | 25 | 193
  White | 75 | 84 | 87 | 33 | 279
  More than one race | 9 | 8 | 10 | 2 | 29
  Unknown or Not Reported | 2 | 3 | 3 | 0 | 8
Care Receiver Marital Status [Count of Participants; unit: Participants]
  Single/Never Married/Partnered | 19 | 18 | 12 | 10 | 59
  Married/Partnered | 57 | 59 | 58 | 24 | 198
  Widowed | 47 | 45 | 49 | 19 | 160
  Separated/Divorced | 21 | 20 | 15 | 9 | 65
  Unknown or Not Reported | 10 | 10 | 20 | 1 | 41
Care Receiver Residence [Count of Participants; unit: Participants]
  Private Home Residence/Adult Group Home | 123 | 115 | 117 | 54 | 409
  Assisted Living Facility/Nursing Home/Skilled Nursing Facility | 18 | 22 | 13 | 2 | 55
  Other | 4 | 5 | 4 | 6 | 19
  Unknown or Not Reported | 9 | 10 | 20 | 1 | 40
Caregiver Distance from Receiver [Count of Participants; unit: Participants]
  With you | 90 | 72 | 81 | 37 | 280
  Less than 1 hour away | 49 | 61 | 42 | 19 | 171
  More than 1 hour away | 4 | 8 | 10 | 6 | 28
  Decline to Answer | 2 | 0 | 1 | 0 | 3
  Unknown or Not Reported | 9 | 11 | 20 | 1 | 41
Caregiver Time Caring [Count of Participants; unit: Participants]
  Less than 1 year | 42 | 46 | 40 | 13 | 141
  1-3 years | 32 | 31 | 28 | 26 | 117
  3 years or more | 69 | 62 | 65 | 22 | 218
  Decline to Answer | 2 | 2 | 1 | 1 | 6
  Unknown or Not Reported | 9 | 11 | 20 | 1 | 41
Caregiver Time Spent Caring per week [Count of Participants; unit: Participants]
  Less than 5 hours | 6 | 10 | 7 | 4 | 27
  5-10 hours | 16 | 20 | 12 | 11 | 59
  11-20 hours | 22 | 13 | 20 | 9 | 64
  More than 20 hours | 100 | 96 | 93 | 37 | 326
  Decline to Answer | 1 | 2 | 2 | 1 | 6
  Unknown or Not Reported | 9 | 11 | 20 | 1 | 41
Caregiver Added Expense [Count of Participants; unit: Participants]
  Yes | 112 | 104 | 100 | 43 | 359
  No | 32 | 36 | 33 | 19 | 120
  Decline to Answer | 1 | 1 | 1 | 0 | 3
  Unknown or Not Reported | 9 | 11 | 20 | 1 | 41
Caregiver Work Status [Count of Participants; unit: Participants]
  Yes | 61 | 66 | 61 | 27 | 215
  No | 83 | 75 | 73 | 35 | 266
  Decline to Answer | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 9 | 11 | 20 | 1 | 41
Caregiver Work Support [Count of Participants; unit: Participants]
  Cut back on hours or quit work entirely | 18 | 15 | 16 | 4 | 53
  Taken an unpaid leave or any leave under Family Medical Leave Act | 5 | 4 | 6 | 1 | 16
  Left one job for a different one | 1 | 3 | 1 | 2 | 7
  Used your own sick leave or vacation time | 20 | 13 | 15 | 9 | 57
  Taken a job or worked additional hours to earn more money | 1 | 0 | 2 | 2 | 5
  None of these apply | 8 | 4 | 6 | 9 | 27
  Decline to Answer | 4 | 8 | 5 | 0 | 17
  Selected More than 1 option | 25 | 29 | 29 | 8 | 91
  Unknown or Not Reported | 72 | 76 | 74 | 28 | 250

OUTCOME MEASURES:

1. Primary Outcome: Table 2. Comparison of 4 Groups
Description: Comparison of 4 groups
  Generalised Anxiety Disorder Assessment (GAD-7) minimum 0 maximum 21 higher scores mean a worse outcome (more anxiety)
  Patient Health Questionnaire 9 (PHQ9) minimum 0 maximum 37 higher scores mean a worse outcome (more distress)
  Caregiver Quality of Life Index (CQLI-R) minimum 0 maximum 40 higher scores mean a better outcome (better quality of life)
Time Frame: from baseline to follow-up (prior to intervention-day 1 to post intervention-approx. day 30)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 (PISCES Face to Face) | Group 2 (PISCES Delivered in a Hybrid Format) | Group 3 (PISCESplus) | Group 4 (PISCESplus Online)
Number analyzed (Participants) | 154 | 152 | 154 | 63
units on a scale
  Difference (FollowUp-Baseline) Generalised Anxiety Disorder Assessment (GAD-7) | -2.54 (4.25) | -1.49 (4.06) | -2.27 (4.56) | -1.52 (5.12)
  Difference (FollowUp-Baseline) Patient Health Questionnaire 9 (PHQ9) | -2.69 (4.29) | -1.56 (4.19) | -1.87 (4.59) | -2.02 (4.14)
  Difference (FollowUp-Baseline) Caregiver Quality of Life Index (CQLI-R) | 1.14 (6.42) | 0.77 (4.82) | 0.27 (7.17) | 1.15 (5.80)
Statistical Analysis 1: Comparison: Group 1 (PISCES Face to Face) vs Group 2 (PISCES Delivered in a Hybrid Format) vs Group 3 (PISCESplus) vs Group 4 (PISCESplus Online); Test type: Other — Group Comparisons; p = 0.1860, Kruskal-Wallis — p-value for Difference (FollowUp-Baseline) Generalised Anxiety Disorder Assessment (GAD-7)
Statistical Analysis 2: Comparison: Group 1 (PISCES Face to Face) vs Group 2 (PISCES Delivered in a Hybrid Format) vs Group 3 (PISCESplus) vs Group 4 (PISCESplus Online); Test type: Other — Group Comparisons; p = 0.2752, Kruskal-Wallis — p-value for Difference (FollowUp-Baseline) Patient Health Questionnaire 9 (PHQ9)
Statistical Analysis 3: Comparison: Group 1 (PISCES Face to Face) vs Group 2 (PISCES Delivered in a Hybrid Format) vs Group 3 (PISCESplus) vs Group 4 (PISCESplus Online); Test type: Other — Group Comparisons; p = 0.6233, Kruskal-Wallis — p-value for Difference (FollowUp-Baseline) Caregiver Quality of Life Index (CQLI-R)

2. Primary Outcome: Table 3. Comparison of Traditional PISCES vs. Online PISCES
Description: Comparison of Traditional PISCES vs. Online PISCES
  Generalised Anxiety Disorder Assessment (GAD-7) minimum 0 maximum 21 higher scores mean a worse outcome (more problems)
  Patient Health Questionnaire 9 (PHQ9) minimum 0 maximum 37 higher scores mean a worse outcome
  Caregiver Quality of Life Index (CQLI-R) minimum 0 maximum 40 higher scores mean a better outcome
Time Frame: from baseline to follow-up (time point 1 is pre-intervention, i.e., day 0 and time point 2 is post-intervention, approx. day 30)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Traditional PISCES: Traditional PISCES
- Online PISCES: Online PISCES
Arm/Group | Traditional PISCES | Online PISCES
Number analyzed (Participants) | 306 | 217
units on a scale
  Difference (FollowUp-Baseline) Generalised Anxiety Disorder Assessment (GAD-7) | -2.04 (4.18) | -2.03 (4.74)
  Difference (FollowUp-Baseline) Patient Health Questionnaire 9 (PHQ9) | -2.15 (4.27) | -1.91 (4.44)
  Difference (FollowUp-Baseline) Caregiver Quality of Life Index (CQLI-R) | 0.96 (5.70) | 0.54 (6.76)
Statistical Analysis 1: Comparison: Traditional PISCES vs Online PISCES; Test type: Other — Group Comparison; p = 0.5638, Wilcoxon (Mann-Whitney) — p-value for Difference (FollowUp-Baseline) Generalised Anxiety Disorder Assessment (GAD-7)
Statistical Analysis 2: Comparison: Traditional PISCES vs Online PISCES; Test type: Other — Group Comparisons; p = 0.9848, Wilcoxon (Mann-Whitney) — p-value for Difference (FollowUp-Baseline) Patient Health Questionnaire 9 (PHQ9)
Statistical Analysis 3: Comparison: Traditional PISCES vs Online PISCES; Test type: Other — Group Comparisons; p = 0.9169, Wilcoxon (Mann-Whitney) — p-value for Difference (FollowUp-Baseline) Caregiver Quality of Life Index (CQLI-R)

3. Primary Outcome: Table 4. Within-Group Comparison Baseline vs. Follow-up
Description: Within-Group Comparison Baseline vs. Follow-up
  Generalised Anxiety Disorder Assessment (GAD-7) minimum 0 maximum 21 higher scores mean a worse outcome (more problems)
  Patient Health Questionnaire 9 (PHQ9) minimum 0 maximum 37 higher scores mean a worse outcome
  Caregiver Quality of Life Index (CQLI-R) minimum 0 maximum 40 higher scores mean a better outcome
Time Frame: from baseline to follow-up (time point 1 is pre-intervention-day 0 and time point 2 is post-intervention-approx. day 30)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Traditional PISCES | Online PISCES
Number analyzed (Participants) | 306 | 217
units on a scale
  Generalised Anxiety Disorder Assessment (GAD-7) | -2.04 (4.18) | -2.03 (4.74)
  Patient Health Questionnaire 9 (PHQ9) | -2.15 (4.27) | -1.91 (4.44)
  Caregiver Quality of Life Index (CQLI-R) | 0.96 (5.70) | 0.54 (6.76)
Statistical Analysis 1: Comparison: Traditional PISCES; Test type: Other — Group Comparisons; p < 0.0001, Wilcoxon Signed Rank Test — p-value for Generalised Anxiety Disorder Assessment (GAD-7) for arm Traditional PISCES
Statistical Analysis 2: Comparison: Traditional PISCES; Test type: Other — Group Comparisons; p < 0.0001, Wilcoxon Signed Rank Test — p-value for Patient Health Questionnaire 9 (PHQ9) for arm Traditional PISCES
Statistical Analysis 3: Comparison: Traditional PISCES; Test type: Other — Group Comparisons; p = 0.0155, Wilcoxon Signed Rank Test — p-value for Caregiver Quality of Life Index (CQLI-R) for arm Traditional PISCES
Statistical Analysis 4: Comparison: Online PISCES; Test type: Other — Group Comparisons; p < 0.0001, Wilcoxon Signed Rank Test — p-value for Generalised Anxiety Disorder Assessment (GAD-7) for arm Online PISCES
Statistical Analysis 5: Comparison: Online PISCES; Test type: Other — Group Comparisons; p < 0.0001, Wilcoxon Signed Rank Test — p-value for Patient Health Questionnaire 9 (PHQ9) for arm Online PISCES
Statistical Analysis 6: Comparison: Online PISCES; Test type: Other — Group Comparisons; p = 0.0504, Wilcoxon Signed Rank Test — p-value for Caregiver Quality of Life Index (CQLI-R) for arm Online PISCES

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the duration of an individual participant's time in the study (which ranged from 4 to 6 weeks).
Description: Given that our intervention was a behavioral intervention with minimal risks. Our definition of adverse event and/or serious adverse event aligns with that of the clinicaltrials.gov Definition.
Arm/Group | Group 1 (PISCES-f2f) | Group 2 (PISCES Video) | Group 3 (PISCESplus) | Group 4 PISCESplus Online
All-Cause Mortality (participants affected / at risk) | 0/154 | 0/152 | 0/154 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/154 | 0/152 | 0/154 | 0/63
Other Adverse Events (participants affected / at risk) | 0/154 | 0/152 | 0/154 | 0/63

LIMITATIONS AND CAVEATS:
Because of the COVID pandemic we implemented some changes in the study protocol for each group and converted data collection to online questionnaires.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT03712410/Prot_SAP_000.pdf